CLINICAL TRIAL: NCT01937689
Title: A Phase I Study of Pyrotinib in Patients With HER2 Positive Advanced Breast Cancer
Brief Title: Study of Pyrotinib in Patients With Human Epidermalgrowth Factor Receptor 2 (HER2) Positive Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLTN-Ib
Record Dates: First submitted 2013-08-14; First posted 2013-09-09 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; advanced; Pyrotinib; Phase I; HER2 positive advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pyrotinib (Experimental): Each subject will receive a single dose of pyrotinib on day 1, followed by 4-day observation period, and then subject will receive pyrotinib once daily for 28 days during cycle 1.Each cycle will consists of 28 days.
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib either at 80, 160, 240, 320, 400, 480 mg ....., p.o. once daily.

SUMMARY:
Pyrotinib is an oral tyrosine kinase inhibitor targeting both HER-1 and HER-2 receptors. This study is designed to evaluate the safety and tolerability of Pyrotinib in patients with HER2 positive advanced breast cancer:

* To evaluate the safety and tolerability of pyrotinib, and the maximum tolerated dose (MTD)
* To determine the dose-limiting toxicity (DLT)
* To determine the pharmacokinetic profile of Pyrotinib and its metabolites
* To assess preliminary antitumor activity
* To determine preliminary regimen dose for phase II study
* To explore the relationship between biomarkers and the toxicity/efficacy of Pyrotinib.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 and ≤70 years.
* ECOG performance status of 0 to 1.
* Life expectancy of more than 12 weeks.
* At least one measurable lesion exists.(RECIST 1.1)
* Histologically or cytologic confirmed HER2 positive advanced breast cancer which failed prior therapies.
* Required laboratory values including following parameters:

  * ANC: ≥ 1.5 x 109/L
  * Platelet count: ≥ 100 x 109/L
  * Hemoglobin: ≥ 9.0 g/dL
  * Total bilirubin: ≤ 1.5 x upper limit of normal, ULN
  * ALT and AST: ≤ 1.5 x ULN
  * BUN and creatine clearance rate: ≥ 50 mL/min
  * LVEF: ≥ 50%
  * QTcF: < 470 ms
* Signed informed consent.

Exclusion Criteria:

* Subjects with third space fluid that can not be controled by drainage or other methods.
* Steroid treatment for more than 50 days, or in need of long-term use of steroids.
* Subjects that are unable to swallow tablets, or dysfunction of gastrointestinal absorption.
* Less than 4 weeks from the last radiotherapy,chemotherapy，surgery，hermone treatment,target therapy, or less than 6 weeks from the nitrosoureas or mitomycin chemotherapy.
* Subjects with uncontrolled hypokalemia and hypomagnesemia before study entry.
* Subjects who can not interrupt the using of the drugs that may cause QT prolongation during study.
* Subjects with intracranial lesions.
* Treated or treating with HER2 tyrosine kinase inhibitors (TKIs) before study entry.
* Receiving any other antitumor therapy.
* Less than 4 weeks from the last clinical trial.
* Known history of hypersensitivity to pyrotinib or any of it components.
* Ongoing infection (determined by investigator).
* History of immunodeficiency, including HIV-positive, suffering from other acquired, congenital immunodeficiency disease, or history of organ transplantation.
* Subjects had any heart disease, including: (1) angina; (2) requiring medication or clinically significant arrhythmia; (3) myocardial infarction; (4) heart failure; (5) Any heart diseases judged by investigator as unsuitable to participate in the trial.
* Female patients who are pregnancy, lactation or women who are of childbearing potential tested positive in baseline pregnancy test.
* Female patients of childbearing age that are reluctant to take effective contraceptive measures throughout the trial period.
* Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study. Examples include, but are not limited to,hypertension, severe diabetes, or thyroid disease.
* Alcoholism, smoking (daily ≥ 5 roots) and other bad habits.
* Known history of neurological or psychiatric disease, including epilepsy or dementia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The maximum-tolerated dose (MTD) will be defined as the maximum dose level at which no more than one subject out of three experiences has a dose-limiting toxicity (DLT) upon completing one treatment cycle. | 4 weeks

SECONDARY OUTCOMES:
Number of participants with adverse events. | 8 weeks
Objective response rate (ORR). | 8 weeks
Pyrotinib pharmacokinetic parameter: Cmax. | 4 weeks
Pyrotinib pharmacokinetic parameter: Tmax. | 4 weeks
Pyrotinib pharmacokinetic parameter: t1/2. | 4 weeks
Pyrotinib pharmacokinetic parameter: AUC. | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Guan X, Ma F, Li Q, Chen S, Lan B, Fan Y, Wang J, Luo Y, Cai R, Zhang P, Li Q, Xu B. Survival benefit and biomarker analysis of pyrotinib or pyrotinib plus capecitabine for patients with HER2-positive metastatic breast cancer: a pooled analysis of two phase I studies. Biomark Res. 2023 Feb 20;11(1):21. doi: 10.1186/s40364-023-00453-0. PMID 36803645
- [Derived] Ma F, Zhu W, Guan Y, Yang L, Xia X, Chen S, Li Q, Guan X, Yi Z, Qian H, Yi X, Xu B. ctDNA dynamics: a novel indicator to track resistance in metastatic breast cancer treated with anti-HER2 therapy. Oncotarget. 2016 Oct 4;7(40):66020-66031. doi: 10.18632/oncotarget.11791. PMID 27602761